CLINICAL TRIAL: NCT00894166
Title: Evaluation of a Tailored Smoking Cessation Treatment Algorithm Based on Initial Treatment Response and Genotype
Acronym: ConNic3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Philip Morris USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00013846
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Results first posted 2012-12-26 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Chantix; varenicline; Nicotine Replacement Therapy; Nicotine Patches; Zyban; bupropion; Quit Smoking
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices; Bupropion; Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Nicotine Replacement Therapy Responder (Active Comparator): Nicotine Responders
  Interventions: Drug: Nicotine Patches
- Pre-Quit Rescue to Bupropion & Nicotine (Active Comparator): Participants not responsive to nicotine patches who are randomly assigned at week 2 to use of Zyban (bupropion) in combination with nicotine patches
  Interventions: Drug: Nicotine patches, then bupropion & nicotine patches (Pre-Quit)
- Pre-Quit Rescue to Varenicline (Active Comparator): Participants not responsive to nicotine patches who are randomly assigned at week 2 to use of Chantix (varenicline)
  Interventions: Drug: Nicotine patches, then varenicline (Pre-Quit)
- Pre-Quit Rescue to Nicotine (Active Comparator): Participants not responsive to nicotine patches who are randomly assigned at week 2 to continued use of nicotine patches
  Interventions: Drug: Nicotine patches, then nicotine patches (Pre-Quit)
- Post-Quit Rescue to Bupropion & Nicotine (Active Comparator): Participants not responsive to nicotine patches who are randomly assigned at week 4 to use of Zyban (bupropion) in combination with nicotine patches
  Interventions: Drug: Nicotine patches, then bupropion & nicotine patches (Post-Quit)
- Post-Quit Rescue to Varenicline (Active Comparator): Participants not responsive to nicotine patches who are randomly assigned at week 4 to use of Chantix (varenicline)
  Interventions: Drug: Nicotine patches, then varenicline (Post-Quit)
- Post-Quit Rescue to Nicotine (Active Comparator): Participants not responsive to nicotine patches who are randomly assigned at week 4 to continued use of nicotine patches
  Interventions: Drug: Nicotine patches, then nicotine patches (Post-Quit)

INTERVENTIONS:
Drug: Nicotine Patches — 21mg (1 patch) or 42mg (2 patches)nicotine patches for first five weeks (# of daily patches based on baseline carbon monoxide level); 21mg nicotine patch for 4 weeks; 14mg nicotine patch for 2 weeks and 7mg nicotine patch for 2 weeks.
  Other Names: NicoDermCQ
  Arms: Nicotine Replacement Therapy Responder
Drug: Nicotine patches, then bupropion & nicotine patches (Pre-Quit) — 21mg (1 patch) or 42mg (2 patches) nicotine patches for first week (# of daily patches based on baseline carbon monoxide level); starting with week 2: 150mg of bupropion once daily and 21mg (1 patch) or 42mg (2 patches)nicotine patches for first 3 days (# of daily patches based on baseline carbon monoxide level); 150mg of bupropion twice daily and 21mg (1 patch) or 42mg (2 patches)nicotine patches for 3 weeks and 4 days (# of daily patches based on baseline carbon monoxide level); 150mg of bupropion twice daily and 21mg nicotine patch for 4 weeks; 150mg of bupropion twice daily and 14mg nicotine patch for 2 weeks and 150mg of bupropion twice daily and 7mg nicotine patch for 2 weeks.
  Other Names: Zyban; NicoDermCQ
  Arms: Pre-Quit Rescue to Bupropion & Nicotine
Drug: Nicotine patches, then varenicline (Pre-Quit) — 21mg (1 patch) or 42mg (2 patches) nicotine patches for first week (# of daily patches based on baseline carbon monoxide level); starting with week 2: 0.5mg of varenicline once daily for first 3 days; 0.5mg of varenicline twice daily for the next 4 days; and 1mg of varenicline twice daily for the remainder of the study (11 weeks)
  Other Names: Chantix; NicoDermCQ
  Arms: Pre-Quit Rescue to Varenicline
Drug: Nicotine patches, then nicotine patches (Pre-Quit) — 21mg (1 patch) or 42mg (2 patches)nicotine patches for first five weeks (# of daily patches based on baseline carbon monoxide level); 21mg nicotine patch for 4 weeks; 14mg nicotine patch for 2 weeks and 7mg nicotine patch for 2 weeks.
  Other Names: NicoDermCQ
  Arms: Pre-Quit Rescue to Nicotine
Drug: Nicotine patches, then bupropion & nicotine patches (Post-Quit) — 21mg (1 patch) or 42mg (2 patches) nicotine patches for first three weeks (# of daily patches based on baseline carbon monoxide level); starting with week 4: 150mg of bupropion once daily and 21mg (1 patch) or 42mg (2 patches) nicotine patches for first 3 days (# of daily patches based on baseline carbon monoxide level); 150mg of bupropion twice daily and 21mg (1 patch) or 42mg (2 patches) nicotine patches for 3 weeks and 4 days (# of daily patches based on baseline carbon monoxide level); 150mg of bupropion twice daily and 21mg nicotine patch for 4 weeks; 150mg of bupropion twice daily and 14mg nicotine patch for 2 weeks and 150mg of bupropion twice daily and 7mg nicotine patch for 2 weeks.
  Other Names: Zyban; NicoDermCQ
  Arms: Post-Quit Rescue to Bupropion & Nicotine
Drug: Nicotine patches, then varenicline (Post-Quit) — 21mg (1 patch) or 42mg (2 patches) nicotine patches for first three weeks (# of daily patches based on baseline carbon monoxide level); starting with week 4: 0.5mg of varenicline once daily for first 3 days; 0.5mg of varenicline twice daily for the next 4 days; and 1mg of varenicline twice daily for the remainder of the study (11 weeks)
  Other Names: Chantix; NicoDermCQ
  Arms: Post-Quit Rescue to Varenicline
Drug: Nicotine patches, then nicotine patches (Post-Quit) — 21mg (1 patch) or 42mg (2 patches) nicotine patches for first seven weeks (# of daily patches based on baseline carbon monoxide level); 21mg nicotine patch for 4 weeks; 14mg nicotine patch for 2 weeks and 7mg nicotine patch for 2 weeks.
  Other Names: NicoDermCQ
  Arms: Post-Quit Rescue to Nicotine

SUMMARY:
Nicotine replacement therapy (NRT) is a well-tolerated and efficacious smoking cessation treatment, and yet many smokers fail to quit using NRT. Many of these smokers may benefit from prescription treatment alternatives, including Zyban or Chantix. In this study, the investigators propose to develop and evaluate a stepped-care treatment algorithm that would evaluate whether smokers who receive treatment with NRT should be supplemented with Zyban or switched to Chantix only based on: 1) their initial response to NRT; and 2) individual genetic factors found to predict smoking cessation in other studies evaluating these treatments. This study is a continuation of our previous studies showing that abstinence rates can be increased by starting nicotine patch therapy two weeks before the quit date. The investigators will provide pre-cessation NRT to all participants initially. Those who do not show a favorable response on early indicators of success (e.g., smoking in the first week after the target quit-smoking date) will receive "rescue" treatment by having their NRT treatment supplemented with Zyban , by being switched to treatment with Chantix or will remain on NRT (control).

The investigators hypothesize that "Rescue" treatment with Zyban in combination with NRT or Chantix will increase success rates over leaving subjects on NRT when they are NRT insufficient responders, i.e. they have shown an unfavorable response to NRT in the first week pre-quit or the first week post-quit.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* smoked an average of at least 10 cigarettes per day for three cumulative years of a brand that delivers (by Federal Trade Commission rated yields) at least 0.5mg nicotine
* expired carbon monoxide reading of at least 15ppm
* express a desire to quit smoking in the next 30 days

Exclusion Criteria:

* Hypertension (systolic >140 mm Hg, diastolic >100 mm Hg, coupled with a history of hypertension); subjects with no previous diagnosis of hypertension may have a screening blood pressure up to 160/100.
* Hypotension (systolic <90 mm Hg, diastolic <60 mm Hg).
* Participants with a history of hypertension may, however, be allowed to participate in the study if the study physician or physician assistant determines that the condition is stable, controlled by medication, and in no way jeopardizes the individual's safety.
* Coronary heart disease;
* Lifetime history of heart attack;
* Cardiac rhythm disorder (irregular heart rhythm);
* Chest pains (unless history, exam, and ECG clearly indicate a non-cardiac source);
* Cardiac (heart) disorder (including but not limited to valvular heart disease, heart murmur, heart failure);
* History of skin allergy;
* Active skin disorder (e.g., psoriasis) within the last five years, except minor skin conditions (including but not limited to facial acne, minor localized infections, and superficial minor wounds);
* Liver or kidney disorder (except kidney stones, gallstones);
* Gastrointestinal problems or disease other than gastroesophageal reflux or heartburn;
* Active ulcers in the past 30 days;
* Lung disorder (including but not limited to Chronic obstructive pulmonary disease (COPD), emphysema, and asthma);
* Brain abnormality (including but not limited to stroke, brain tumor, and seizure disorder);
* History of migraine headaches in the past 5 years;
* History of fainting;
* Problems giving blood samples;
* Diabetes treated with insulin; non-insulin treated diabetes (unless glucose is less than 180mg/dcl and HbA1c is less than 7%);
* Current cancer or treatment for cancer in the past six months (except basal or squamous cell skin cancer);
* Other major medical condition;
* Current psychiatric disease (with the exception of anxiety disorders, Obsessive-compulsive disorder (OCD) and ADHD);
* Suicidal ideation (within the past 10 years) or lifetime occurrence of attempted suicide;
* Current depression - The Patient Health Questionnaire (PHQ-9) for Depression will be used to screen for current (within 2 weeks) depression. Potential subjects who score >9 (or who score >0 on item #9 ("Thoughts that you would be better off dead, or of hurting yourself in some way") will be excluded from study participation, and, at the discretion of the study physician, referred to appropriate psychiatric treatment;
* Bulimia or anorexia;
* Pregnant or nursing mothers;
* Use (within the past 30 days) of:
* Illegal drugs (or if the urine drug screen is positive),
* Experimental (investigational) drugs;
* Psychiatric medications including antidepressants, anti-psychotics or any other medications that are known to affect smoking cessation (e.g. clonidine);
* Opiate medications for pain or sleep (non-opiate medication for pain or sleep will be allowed)
* Smokeless tobacco (chewing tobacco, snuff), cigars or pipes;
* Wellbutrin, bupropion, Zyban, Chantix, nicotine replacement therapy or any other smoking cessation aid.
* Alcohol abuse - The AUDIT (Alcohol Use Disorders Identification Test) questionnaire will be used to assess alcohol abuse. Potential participants will be asked the first two questions on the AUDIT questionnaire during the phone screen. If the person scores "4" on both questions, a screening appointment will not be scheduled. During the screening session the entire AUDIT questionnaire will be administered. Females who score greater than or equal to 13 and males who score greater than or equal to 15 will be excluded from the study.
* Significant adverse reaction to Wellbutrin / Zyban or Chantix / Varenicline in the past

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jed E Rose, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke Center for Nicotine & Smoking Cessation Research, Charlotte, Durham, Raleigh, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Rose JE, Behm FM. Adapting smoking cessation treatment according to initial response to precessation nicotine patch. Am J Psychiatry. 2013 Aug;170(8):860-7. doi: 10.1176/appi.ajp.2013.12070919. PMID 23640009
- [Derived] Uhl GR, Walther D, Musci R, Fisher C, Anthony JC, Storr CL, Behm FM, Eaton WW, Ialongo N, Rose JE. Smoking quit success genotype score predicts quit success and distinct patterns of developmental involvement with common addictive substances. Mol Psychiatry. 2014 Jan;19(1):50-4. doi: 10.1038/mp.2012.155. Epub 2012 Nov 6. PMID 23128154

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study started June 2009 and ended April 2011 and was conducted at Duke University Medical Center.
Pre-assignment Details: All enrollees began nicotine patches & those who didn't show a >50% reduction in expired air carbon monoxide (CO) at 1 week (1 week before the target quit date) or who lapsed in the 1st week after their quit date were randomized to one of 6 groups. The 7th group - Nicotine Replacement Therapy (NRT) Responders were excluded from this randomization.
Groups:
- NRT Responder: Participants in this group showed both a >50% decrease in expired air CO during the 1st week of pre-cessation nicotine patch treatment and did not lapse during their 1st week after quitting.
  21mg (1 patch) or 42mg (2 patches)nicotine patches for first five weeks (# of daily patches based on baseline carbon monoxide level); 21mg nicotine patch for 4 weeks; 14mg nicotine patch for 2 weeks and 7mg nicotine patch for 2 weeks.
- Pre-Quit Randomization to Bupropion + NRT: Participants not showing a >50% decrease in expired air CO during the 1st week of pre-cessation nicotine patch treatment, who are randomly assigned at week 2 to use Zyban (bupropion) in combination with nicotine patches.
  21mg (1 patch) or 42mg (2 patches) nicotine patches for first week (# of daily patches based on baseline carbon monoxide level); starting with week 2: 150mg of bupropion once daily and 21mg (1 patch) or 42mg (2 patches)nicotine patches for first 3 days (# of daily patches based on baseline carbon monoxide level); 150mg of bupropion twice daily and 21mg (1 patch) or 42mg (2 patches)nicotine patches for 3 weeks and 4 days (# of daily patches based on baseline carbon monoxide level); 150mg of bupropion twice daily and 21mg nicotine patch for 4 weeks; 150mg of bupropion twice daily and 14mg nicotine patch for 2 weeks and 150mg of bupropion twice daily and 7mg nicotine patch for 2 weeks.
- Pre-Quit Randomization to Varenicline: Participants not showing a >50% decrease in expired air CO during the 1st week of pre-cessation nicotine patch treatment, who are randomly assigned at week 2 to use varenicline.
  21mg (1 patch) or 42mg (2 patches) nicotine patches for first week (# of daily patches based on baseline carbon monoxide level); starting with week 2: 0.5mg of varenicline once daily for first 3 days; 0.5mg of varenicline twice daily for the next 4 days; and 1mg of varenicline twice daily for the remainder of the study (11 weeks).
- Pre-Quit Randomization to NRT: Participants not showing a >50% decrease in expired air CO during the 1st week of pre-cessation nicotine patch treatment,who are randomly assigned at week 2 to use continued use of nicotine patches.
  21mg (1 patch) or 42mg (2 patches)nicotine patches for first five weeks (# of daily patches based on baseline carbon monoxide level); 21mg nicotine patch for 4 weeks; 14mg nicotine patch for 2 weeks and 7mg nicotine patch for 2 weeks.
- Post-Quit Randomization to Bupropion + NRT: Participants who did show >50% decrease in expired air CO on pre-cessation NRT but who lapsed during the first week post quit date, who are randomly assigned to use of bupropion in combination with nicotine patches.
  21mg (1 patch) or 42mg (2 patches) nicotine patches for first three weeks (# of daily patches based on baseline carbon monoxide level); starting with week 4: 150mg of bupropion once daily and 21mg (1 patch) or 42mg (2 patches) nicotine patches for first 3 days (# of daily patches based on baseline carbon monoxide level); 150mg of bupropion twice daily and 21mg (1 patch) or 42mg (2 patches) nicotine patches for 3 weeks and 4 days (# of daily patches based on baseline carbon monoxide level); 150mg of bupropion twice daily and 21mg nicotine patch for 4 weeks; 150mg of bupropion twice daily and 14mg nicotine patch for 2 weeks and 150mg of bupropion twice daily and 7mg nicotine patch for 2 weeks.
- Post-Quit Randomized to Varenicline: Participants who did show >50% decrease in expired air CO on pre-cessation NRT but who lapsed during the first week post quit date, who are randomly assigned to use varenicline.
  21mg (1 patch) or 42mg (2 patches) nicotine patches for first three weeks (# of daily patches based on baseline carbon monoxide level); starting with week 4: 0.5mg of varenicline once daily for first 3 days; 0.5mg of varenicline twice daily for the next 4 days; and 1mg of varenicline twice daily for the remainder of the study (11 weeks).
- Post-Quit Randomized to NRT: Participants who did show >50% decrease in expired air CO on pre-cessation NRT but who lapsed during the first week post quit date, who are randomly assigned to use nicotine patches.
  21mg (1 patch) or 42mg (2 patches) nicotine patches for first seven weeks (# of daily patches based on baseline carbon monoxide level); 21mg nicotine patch for 4 weeks; 14mg nicotine patch for 2 weeks and 7mg nicotine patch for 2 weeks.
- Withdrew Prior to Randomization: These subjects dropped from study participation after the first study session; therefore, they were never randomized into one of the study groups.
  21mg (1 patch) or 42mg (2 patches) nicotine patches were dispensed for the first week of study participation during the one session they completed.
Period: Overall Study
Arm/Group | NRT Responder | Pre-Quit Randomization to Bupropion + NRT | Pre-Quit Randomization to Varenicline | Pre-Quit Randomization to NRT | Post-Quit Randomization to Bupropion + NRT | Post-Quit Randomized to Varenicline | Post-Quit Randomized to NRT | Withdrew Prior to Randomization
Started | 132 | 109 | 112 | 114 | 34 | 36 | 35 | 34
Completed | 71 | 46 | 50 | 45 | 10 | 20 | 19 | 0
Not Completed | 61 | 63 | 62 | 69 | 24 | 16 | 16 | 34
Not completed — Withdrew or Lost to Follow-Up | 61 | 63 | 62 | 68 | 24 | 16 | 16 | 34
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- NRT Responder: Participants in this group showed both a >50% decrease in expired air CO during the 1st week of pre-cessation nicotine patch treatment and did not lapse during their 1st week after quitting.
- Pre-Quit Randomization to Bupropion + NRT: Participants not showing a >50% decrease in expired air CO during the 1st week of pre-cessation nicotine patch treatment, who are randomly assigned at week 2 to use Zyban (bupropion) in combination with nicotine patches.
- Pre-Quit Randomization to Varenicline: Participants not showing a >50% decrease in expired air CO during the 1st week of pre-cessation nicotine patch treatment, who are randomly assigned at week 2 to use varenicline.
- Pre-Quit Randomization to NRT: Participants not showing a >50% decrease in expired air CO during the 1st week of pre-cessation nicotine patch treatment,who are randomly assigned at week 2 to use continued use of nicotine patches.
- Post-Quit Randomization to Bupropion + NRT: Participants who did show >50% decrease in expired air CO on pre-cessation NRT but who lapsed during the first week post quit date, who are randomly assigned to use of bupropion in combination with nicotine patches.
- Post-Quit Randomized to Varenicline: Participants who did show >50% decrease in expired air CO on pre-cessation NRT but who lapsed during the first week post quit date, who are randomly assigned to use varenicline.
- Post-Quit Randomized to NRT: Participants who did show >50% decrease in expired air CO on pre-cessation NRT but who lapsed during the first week post quit date, who are randomly assigned to use nicotine patches.
- Withdrew Prior to Randomization: These subjects dropped from study participation after the first study session; therefore, they were never randomized into one of the study groups.
- Total: Total of all reporting groups
Arm/Group | NRT Responder | Pre-Quit Randomization to Bupropion + NRT | Pre-Quit Randomization to Varenicline | Pre-Quit Randomization to NRT | Post-Quit Randomization to Bupropion + NRT | Post-Quit Randomized to Varenicline | Post-Quit Randomized to NRT | Withdrew Prior to Randomization | Total
Number analyzed (Participants) | 132 | 109 | 112 | 114 | 34 | 36 | 35 | 34 | 606
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 129 | 108 | 112 | 113 | 34 | 36 | 35 | 34 | 601
  >=65 years | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 43.6 (10.2) | 46.0 (10.8) | 44.7 (10.7) | 44.3 (10.8) | 43.1 (11.6) | 44.1 (11.2) | 40.8 (12.8) | 40.7 (10.1) | 44.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 50 | 49 | 61 | 17 | 17 | 22 | 16 | 300
  Male | 64 | 59 | 63 | 53 | 17 | 19 | 13 | 18 | 306
Region of Enrollment [Number; unit: participants]
  United States | 132 | 109 | 112 | 114 | 34 | 36 | 35 | 34 | 606

OUTCOME MEASURES:

1. Primary Outcome: Continuous 4-week Abstinence From Smoking Between Weeks 8-11 After the Quit Date (Through the End of Treatment)
Description: A self report of no cigarettes smoked confirmed by expired air carbon monoxide of <=10ppm was the criterion for abstinence.
Time Frame: weeks 8-11 after quit date
Population: All participants were included in the analyses except those dropping out prior to randomization points, those censored for taking contraindicated medications or failing to meet other inclusion criteria, and one death having no apparent relationship to treatment.
Measure: Number (95% Confidence Interval); unit: percentage of subjects abstinent
Arm/Group | NRT Responder | Pre-Quit Randomization to Bupropion + NRT | Pre-Quit Randomization to Varenicline | Pre-Quit Randomization to NRT | Post-Quit Randomization to Bupropion + NRT | Post-Quit Randomized to Varenicline | Post-Quit Randomized to NRT
Number analyzed (Participants) | 120 | 99 | 103 | 106 | 30 | 35 | 30
percentage of subjects abstinent | 59.2 [50.4 to 68] | 28.3 [19.4 to 37.2] | 23.3 [15.1 to 31.5] | 16.0 [9 to 23] | 26.7 [10.9 to 42.5] | 37.1 [21.1 to 53.1] | 26.7 [10.9 to 42.5]

2. Secondary Outcome: Abstinence (7 Days) at 6 Months.
Time Frame: point abstinence (7 days) at 6 months post-quit date
Measure: Number; unit: percentage of subjects
Arm/Group | NRT Responder | Pre-Quit Randomization to Bupropion + NRT | Pre-Quit Randomization to Varenicline | Pre-Quit Randomization to NRT | Post-Quit Randomization to Bupropion + NRT | Post-Quit Randomized to Varenicline | Post-Quit Randomized to NRT
Number analyzed (Participants) | 120 | 99 | 108 | 106 | 30 | 35 | 30
percentage of subjects | 21.7 | 17.2 | 16.5 | 6.6 | 10.0 | 20.0 | 13.3

3. Secondary Outcome: Continuous Abstinence From Smoking at 6 Months Post Quit.
Time Frame: continuous abstinence at 6 months post quit day
Measure: Number; unit: percentage of subjects
Arm/Group | NRT Responder | Pre-Quit Randomization to Bupropion + NRT | Pre-Quit Randomization to Varenicline | Pre-Quit Randomization to NRT | Post-Quit Randomization to Bupropion + NRT | Post-Quit Randomized to Varenicline | Post-Quit Randomized to NRT
Number analyzed (Participants) | 120 | 99 | 108 | 106 | 30 | 35 | 30
percentage of subjects | 20.0 | 13.1 | 5.8 | 5.8 | 10.0 | 14.3 | 10.0

ADVERSE EVENTS:
Time Frame: Subjects were receiving study drugs for 11-13 weeks. At each study session during this period subjects completed a questionnaire about side effects. Subjects were also told to contact us between study sessions if side effects were bothersome.
Description: 34 subjects withdrew from participation prior to Session P2 and were therefore not randomized into one of the study groups. These participates received nicotine patches for the first week of the study but did not attend the second session so no data about adverse events were collected.
Arm/Group | NRT Responder | Pre-Quit Randomization to Bupropion + NRT | Pre-Quit Randomization to Varenicline | Pre-Quit Randomization to NRT | Post-Quit Randomization to Bupropion + NRT | Post-Quit Randomized to Varenicline | Post-Quit Randomized to NRT
Serious Adverse Events (participants affected / at risk) | 3/132 | 4/109 | 3/112 | 2/114 | 2/34 | 1/36 | 1/35
Other Adverse Events (participants affected / at risk) | 88/132 | 74/109 | 64/112 | 85/114 | 31/34 | 27/36 | 28/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NRT Responder (N=132) | Pre-Quit Randomization to Bupropion + NRT (N=109) | Pre-Quit Randomization to Varenicline (N=112) | Pre-Quit Randomization to NRT (N=114) | Post-Quit Randomization to Bupropion + NRT (N=34) | Post-Quit Randomized to Varenicline (N=36) | Post-Quit Randomized to NRT (N=35)
Chest Pain, shortness of breath, vision loss (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hives, itching, knot in throat (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain, myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain worsened with inspiration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
psychiatric side effects (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
urticaria and shortness of breath (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
paroxsymal supraventricular tachycardia and fainting (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
chest pain, new left bundle branch block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain, unifocal PVCs (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash distant from patch site (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucinations, chest pains, vomiting (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body aches, generalized weakness, sensation of throat swelling, lightheadedness,difficulty breathing (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
stroke and death (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
myocardial infaction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NRT Responder (N=132) | Pre-Quit Randomization to Bupropion + NRT (N=109) | Pre-Quit Randomization to Varenicline (N=112) | Pre-Quit Randomization to NRT (N=114) | Post-Quit Randomization to Bupropion + NRT (N=34) | Post-Quit Randomized to Varenicline (N=36) | Post-Quit Randomized to NRT (N=35)
HEADACHE (Nervous system disorders) | 18 (23) | 17 (21) | 9 (9) | 17 (22) | 5 (11) | 6 (7) | 4 (11)
EXCESSIVE SWEATING (General disorders) | 7 (8) | 12 (21) | 4 (5) | 12 (18) | 4 (4) | 3 (6) | 6 (8)
SWELLING (General disorders) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
MOUTH/THROAT IRRITATION (General disorders) | 11 (15) | 7 (9) | 2 (2) | 4 (6) | 2 (4) | 1 (1) | 4 (4)
DRY MOUTH (General disorders) | 14 (24) | 19 (43) | 7 (14) | 18 (28) | 8 (22) | 4 (7) | 8 (25)
THIRST (General disorders) | 19 (33) | 21 (41) | 12 (25) | 23 (36) | 10 (24) | 8 (12) | 8 (25)
COUGHING (Respiratory, thoracic and mediastinal disorders) | 10 (16) | 11 (21) | 15 (29) | 13 (17) | 4 (9) | 5 (6) | 6 (8)
CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
JOINT / MUSCLE PAIN (Musculoskeletal and connective tissue disorders) | 14 (22) | 4 (6) | 4 (7) | 9 (10) | 7 (19) | 3 (5) | 4 (10)
HEARTBURN (Gastrointestinal disorders) | 9 (11) | 7 (18) | 4 (7) | 4 (6) | 4 (11) | 3 (4) | 2 (3)
NAUSEA (Gastrointestinal disorders) | 9 (11) | 4 (4) | 4 (5) | 4 (4) | 4 (5) | 3 (4) | 3 (4)
CONSTIPATION (Gastrointestinal disorders) | 7 (13) | 9 (16) | 3 (3) | 6 (9) | 1 (3) | 2 (2) | 4 (13)
UPSET STOMACH (Gastrointestinal disorders) | 8 (8) | 3 (3) | 3 (5) | 6 (8) | 2 (3) | 1 (1) | 2 (3)
DIARRHEA (Gastrointestinal disorders) | 1 (1) | 2 (3) | 6 (7) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
IRRITABILITY (Nervous system disorders) | 20 (35) | 16 (22) | 18 (31) | 15 (31) | 9 (15) | 12 (22) | 7 (10)
NIGHTMARES (Nervous system disorders) | 8 (11) | 5 (8) | 8 (8) | 9 (9) | 0 (0) | 1 (1) | 7 (10)
VIVID DREAMS (Nervous system disorders) | 36 (85) | 35 (74) | 25 (50) | 39 (87) | 12 (38) | 14 (28) | 17 (51)
INSOMNIA (Nervous system disorders) | 20 (33) | 26 (37) | 14 (17) | 20 (34) | 11 (29) | 6 (16) | 9 (14)
DEPRESSION (Psychiatric disorders) | 3 (6) | 3 (3) | 6 (8) | 8 (11) | 0 (0) | 2 (3) | 3 (4)
ANXIETY (Psychiatric disorders) | 14 (15) | 16 (26) | 8 (15) | 9 (23) | 6 (10) | 2 (5) | 7 (9)
TREMOR (Nervous system disorders) | 1 (1) | 5 (6) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
DECREASED LIBIDO (Nervous system disorders) | 5 (5) | 4 (10) | 6 (12) | 2 (6) | 1 (1) | 0 (0) | 1 (1)
ITCHING/BURNING AT PATCH SITE (Skin and subcutaneous tissue disorders) | 27 (63) | 19 (28) | 13 (14) | 30 (44) | 10 (26) | 7 (11) | 11 (26)
RASH AT PATCH SITE (Skin and subcutaneous tissue disorders) | 17 (30) | 8 (9) | 6 (7) | 10 (15) | 2 (4) | 3 (3) | 6 (12)
RASH DISTANT FROM PATCH SITE (General disorders) | 4 (6) | 3 (3) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The group sizes for the post quit date randomization groups was relatively small. Second, the study used a tailored dose of pre-cessation nicotine patch therapy that is not in accordance with current product labeling in the US.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No